CLINICAL TRIAL: NCT02177084
Title: Percutaneous Tibial Nerve Stimulation in the Treatment of Anterior Resection Syndrome After Rectal Cancer Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Cuicchi Dajana, Dr Dajana Cuicchi MD PhD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTNS BO-01
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Rectal Cancer; Low Anterior Resection Syndrome
Keywords: PTNS; rectal cancer; low anterior resection syndrome
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome

ARMS (2):
- PTNS + conservative treatment (Experimental): PTNS consists in the insertion of a small electrode above the medial malleolus adjacent to the posterior tibial nerve. An adhesive surface electrode is placed under th arch of the foot. Both electrodes are connected to the neurostimulator that generates electricity. A neuromodulation session lasts 30 minutes.
  The treatment plan includes 12 weekly sessions, followed by two sessions at 2-week intervals and the last one after one month. Two additional sessions of reinforcement (top-up) are provided at intervals of 6 months or earlier in case of worsening of symptoms
  Interventions: Device: PTNS
- conservative treatment (No Intervention)

INTERVENTIONS:
Device: PTNS
  Arms: PTNS + conservative treatment

SUMMARY:
The study aims to evaluate the efficacy of percutaneous tibial nerve stimulation (PTNS) associated with conservative therapy (arm A) for the treatment of low anterior resection syndrome (LARS) compared with only conservative therapy (arm B).

The secondary aims are the evaluation of the following parameters:

* Effect of PTNS on manometric parameters
* Effect of PTNS on quality of life
* Effect of PTNS on the severity of fecal incontinence and / or obstructed defecation
* Safety of PTNS

DETAILED DESCRIPTION:
The study is a prospective randomized clinical trial that compares two treatments in patients with LARS:

Arm A: PTNS + conservative treatment (based on predominant symptom) Arm B: only conservative treatment

The study is divided into two phases:

1. PRETREATMENT PHASE

   The patients with LARS score ≥ 21 after anterior resection of the rectum with sphincter-saving surgery for rectal cancer, will be submitted during the first visit of the study to :
   * Collection of personal data
   * Collection of medical records
   * Collection of data relating to the intervention of anterior resection of the rectum
   * Verification of the criteria for inclusion / exclusion
   * Collection of informed consent
   * Administration of the questionnaires European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Cancer 30 (EORTC QLQ-C30), European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire Colorectal 38 (EORTC QLQ-CR38), Faecal incontinence severity index (FISI); Fecal incontinence quality of life questionnaire (FIQL), Obstructed defaecation syndrome (ODS) score questionnaire and Constipation-related quality of life questionnaire (CRQoL)
   * Endoanal ultrasound
   * Anorectal manometry
2. PHASE OF TREATMENT During the treatment phase, data related to the treatment and any treatment related-complications will be recorded on a special form Bowel function and quality of life will be assessed using the same questionnaires at the end of treatment. Even anorectal manometry will be repeated at the end of treatment.

It is expected to enroll approximately 12 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LARS score ≥ 21 after anterior resection of the rectum with sphincter-saving surgery for rectal cancer;
* Age> 18 years;
* Obtaining informed consent.

Exclusion Criteria:

* Patients carrying ostomy;
* Patients with clinical or radiological evidence of local or distant tumor recurrence;
* Patients suffering from neurological disorders;
* Patients with Inflammatory Bowel Disease (IBD);
* Patients who have a pacemaker or defibrillator;
* Patients taking antiplatelet agents or anticoagulants;
* Patients unable to follow the procedures of the Protocol or to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
LARS score | 67 weeks
  The primary end point is the evaluation of the results of the two interventions in functional terms, by comparing the LARS score calculated first at the end and after 12 months of treatment, according to the following classification:
  * No LARS: a score between 0 and 20
  * LARS mild: score between 21:29
  * LARS severe: a score between 30 and 42

SECONDARY OUTCOMES:
EORTC QLQ-CR38 | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires EORTC QLQ-CR38 performed before and after treatment.
EORTC QLQ-C30 | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires EORTC QLQ-C30 performed before and after treatment
FISI | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires FISI examinations performed before and after treatment.
FIQL | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires FIQL performed before and after treatment.
ODS SCORE | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires ODS score performed before and after treatment.
CRQoL | 67 weeks
  Secondary objectives will be evaluated by the change of the questionnaires CRQoL performed before and after treatment.
functional outcome | 67 weeks
  Functional outcome will be evaluated comparing manometric examinations performed before and after treatment.
morbidity | 67 weeks
  registration of complications after each therapy session

CONTACTS AND LOCATIONS:
Locations (1):
- S'Orsola Malpighi University Hospital, Bologna, Bologna, Italy